CLINICAL TRIAL: NCT00510900
Title: Effects of Left Atrial Appendage Occlusion
Status: Withdrawn | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 0508103
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The proposed work seeks to further understand the effects of LAA occlusion on cardiac structure and function, and in homeostasis.

Numerous studies have implicated the left atrial appendage (LAA) as the source of the vast majority of left atrial thrombi in the setting of AF3.

The University of Pittsburgh Medical Center will be implanting a Left Atrial Appendage filter system (the WATCHMAN® Left Atrial Appendage Filter System, manufactured by Atritech, Inc.). We aim to follow these patients for six months post implant in order to assess their heart rhythm, function, and to do blood tests to evaluate for neurohormonal changes.

DETAILED DESCRIPTION:
Atrial fibrillation (AF), a heart rhythm disorder, is a major health problem. As many as 3 million US persons are afflicted; this number is expected to rise significantly in coming decades because AF incidence is directly correlated with age1. AF is significantly associated with cardiovascular morbidity and mortality.

The University of Pittsburgh Medical Center will be implanting a Left Atrial Appendage filter system (the WATCHMAN® Left Atrial Appendage Filter System, manufactured by Atritech, Inc.). We aim to follow these patients for six months post implant in order to assess:

1. Blood tests to monitor biochemical markers of cardiac remodeling and indices of heart function. We will assess atrial natriuretic factor; brain natriuretic peptide; norepinephrine; matrix metalloproteinases 1, 2, 3, 8, 9, and 13; gelatinases 2 and 9; soluble tumor necrotic factor-II; angiotensin; aldosterone; ADH; rennin; interleukin-6; TNF-α; homocysteine; C-reactive protein; quantitative D-dimer; fibrin; fibrinogen; and fibrin split products. Biochemical markers of cardiac remodeling are being intensively studied globally, with novel markers discovered and published frequently. Serum will be banked for the duration of the study to allow for retrospective investigation of newly published markers.
2. Echocardiogram to evaluate myocardial function and atrial work.
3. 24 hour holter monitor to evaluate the subjects' heart rhythm for presence or absence of atrial fibrillation.

This study will be a non-blinded observational study with a control group. Subjects will be recruited from the patient pool of the Principal Investigator and Co-Investigators. All subjects in the intervention group will have had the WATCHMAN device implanted at UPMC. The control group in this trial will be comprised of age-matched controls from the control group in the WATCHMAN device trial, also from the patient pool of the Principal Investigator and Co-Investigators. Subjects will be approached by one of the Investigators.

The primary outcome of interest will be left atrial work, measured on a continuous scale. Analysis of covariance (ANCOVA) will be used to compare mean left atrial work scores at 12 months between the intervention and non-intervention patient groups adjusting for baseline values.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Ability to give informed consent.
* Patient will be enrolled in the WATCHMAN device trial at UPMC. 4 -Documented history of atrial fibrillation.

Exclusion Criteria:

* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Schwartzman, MD, Principal Investigator — University of Pittsburgh/UPMC
Locations (1):
- University of Pittsburgh Medical Center/Comprehensive Heart Ctr., Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Background] Furberg CD, Psaty BM, Manolio TA, Gardin JM, Smith VE, Rautaharju PM. Prevalence of atrial fibrillation in elderly subjects (the Cardiovascular Health Study). Am J Cardiol. 1994 Aug 1;74(3):236-41. doi: 10.1016/0002-9149(94)90363-8. PMID 8037127
- [Background] Al-Saady NM, Obel OA, Camm AJ. Left atrial appendage: structure, function, and role in thromboembolism. Heart. 1999 Nov;82(5):547-54. doi: 10.1136/hrt.82.5.547. PMID 10525506